CLINICAL TRIAL: NCT00869180
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of a Diclofenac Sodium Patch for the Topical Treatment of Acute Pain Due to Mild to Moderate Ankle Sprain
Brief Title: Diclofenac Patch for Treatment of Acute Pain Due to Mild to Moderate Ankle Sprain
Acronym: SUPPORT 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cerimon Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Shaily J. Reichert, V.P. of Clinical Development, Cerimon Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCF-004
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Acute Pain; Ankle Sprain
Keywords: diclofenac; ankle sprain; acute pain; topical; patch; Acute Pain due to Mild to Moderate Ankle Sprain
MeSH Terms: conditions — Acute Pain; Ankle Injuries | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac Sodium Patch (Experimental)
  Interventions: Drug: Diclofenac Sodium
- Topical Placebo Patch (Placebo Comparator)
  Interventions: Drug: Matching Placebo Patch

INTERVENTIONS:
Drug: Diclofenac Sodium — Topical diclofenac patch applied once daily to area of pain
  Arms: Diclofenac Sodium Patch
Drug: Matching Placebo Patch — Matching placebo patch, containing identical constituents to the active comparator except for diclofenac sodium; applied once daily
  Arms: Topical Placebo Patch

SUMMARY:
The primary purpose of this study is to assess the effectiveness of once daily application of a diclofenac sodium topical patch in reducing acute pain due to mild to moderate ankle sprains when applied to the painful area.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, parallel group study will be conducted in patients with mild or moderate ankle sprains.

Eligible patients will be randomized (in a 1:1 ratio) to receive double-blind treatment with either the diclofenac topical patch or a matching placebo patch to be applied once daily for 7 days. Patients will return to the clinic for assessments on Day 3 and Day 7; a follow-up assessment will be conducted on Day 14. Patients will complete an electronic diary in which assessments including pain intensity, pain relief and functional disability will be recorded twice daily. Ratings of the quality of sleep will be recorded in the diary each morning, and the use of study treatment and rescue medication will be recorded in the diary each day.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 17 - 75 years of age
* Sustained recent, painful unilateral mild to moderate ankle sprain
* Meet baseline pain criterion

Exclusion Criteria:

* Open wound or infection at site of injury
* Evidence of severe injury or ankle fracture
* Use of oral NSAIDs or opioids within 12 - 24 hours of injury
* Presence or history of peptic ulcers or GI bleeding
* A history of intolerance to NSAIDs, acetaminophen, adhesives
* Positive pregnancy test
* Positive drug screen

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in average pain during daily activity at Day 3 | Day 3

SECONDARY OUTCOMES:
Change in average pain during daily activity at Day 7 | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States